CLINICAL TRIAL: NCT02219035
Title: A Prospective Investigation of the VWF-ADAMTS 13 Axis in Acute Ischaemic Brain Injury (TIAs and Stroke).
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 14/0088
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Stroke
Keywords: presentation with
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- stroke-ischaemic: no interventions
- stroke -haemorrhagic: no intervention
- stroke: not confirmed: no intervention

SUMMARY:
In patients presenting with acute stroke or transient ischaemic attacks (TIA), von Willebrand factor related parameters, including VWF antigen, activity, FVIII:c and propeptides, ADAMTS13 levels and VWF multimers in cases where ADAMTS 13 was reduced will be measured. Global haemostasis will be assessed using thrombin generation and the relation between increase thrombin generation and VWF explored. Thrombin generation will be performed pre and post filtration for the presence of procoagulant microparticles. These parameters will be investigated acutely, at presentation and in convalescence; in addition, the effect on these parameters of treatment such as thrombolysis may be informative. Correlation between measured parameters and adverse clinical outcome would be used to identify markers of severity and progression of ischaemic stroke and identification of potential novel approaches to therapy that might improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years of age presenting within 9 hours of onset of symptoms will be recruited from the hyperacute stroke unit at UCLH.
* Patients in whom stroke has been excluded or in whom intracerebral haemorrhage has been diagnosed are to be included as 'controls'. The definitive diagnosis will not be immediately obvious at presentation.
* Written consent will be obtained from patients or their nearest relative, particularly in patients with aphasia/dysphasia.

Exclusion Criteria:

* Patients <18 years old
* Patients with systemic vasculitis or active malignancy will be excluded.
* Patients not wishing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all acute admissions presenting with ? stroke
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Acute ischemic stroke/TIAs are associated with increased levels and activity of VWF and low levels of ADAMTS13 activity. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie Scully, Principal Investigator — UCLH
Locations (1):
- UCLH, London, United Kingdom